CLINICAL TRIAL: NCT00973479
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial of Golimumab, an Anti-TNFalpha Monoclonal Antibody, Administered Intravenously, in Patients With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Brief Title: An Effectiveness and Safety Study of Intravenous Golimumab in Patients With Active Rheumatoid Arthritis Despite Treatment With Methotrexate Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR015784; CNTO148ART3001 (Other: Centocor, Inc); 2008-006064-11 (EudraCT Number)
Record Dates: First submitted 2009-09-04; First posted 2009-09-09 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, Rheumatoid; Active rheumatoid arthritis; Golimumab; CNTO148; Anti-TNFalpha monoclonal antibody; Methotrexate; Intravenous
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — golimumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I: Placebo + Methotrexate (MTX) (Experimental): Participants will receive placebo at Weeks 0, 4, 12, and 16. Participants will cross over to golimumab at Week 24, and receive administrations at Weeks 24, 28, and every 8 weeks thereafter. They will be maintained on their stable dose of commercial methotrexate throughout the study. Participants will be eligible for early escape (receive golimumab) at Week 16 if they demonstrate a less than 10 percent improvement in both tender and swollen joint count. These participants will receive golimumab at Weeks 16, 20, and every 8 weeks thereafter.
  Interventions: Drug: Golimumab; Other: Placebo; Drug: methotrexate (MTX)
- Group II: Golimumab + Methotrexate (MTX) (Placebo Comparator): Participants will receive golimumab at Weeks 0, 4, and every 8 weeks thereafter. They will be maintained on their stable dose of commercial methotrexate throughout the study. Participants will receive a placebo infusion at Week 16 and Week 24 to maintain the blind.
  Interventions: Drug: Golimumab; Other: Placebo; Drug: methotrexate (MTX)

INTERVENTIONS:
Drug: Golimumab — Participants will receive 2 mg/kg of golimumab intravenously over 30 ± 10 minutes. Group 1: at Weeks 0, 4, and every 8 weeks thereafter (up to Week 100). Group II: Weeks 24, 28, and every 8 weeks thereafter (up to Week 100); Early escape: at Week 16, 20 and every 8 weeks thereafter (up to Week 100).
Other: Placebo — Participants will receive placebo intravenous infusion over 30 ± 10 minutes as: Group I: at Week 16 and 24; Group II: at Weeks 0, 4, 12, 16, and 20; and for early escape: at Week 24.
Drug: methotrexate (MTX) — Participants will be maintained on their stable dose of commercial MTX (between 15 to 25 mg/week) throughout the study.

SUMMARY:
The purpose of this study is to evaluate clinical effectiveness and safety of golimumab with methotrexate (MTX) in the treatment of rheumatoid arthritis (RA) when compared to MTX alone.

DETAILED DESCRIPTION:
This is a randomized (study medication is assigned by chance), double-blind (neither physician nor participants knows the treatment that the participant receives), placebo-controlled (an inactive substance is compared with a medication to test whether the medication has a real effect in a clinical study), multicenter, 2-arm (2 groups) study of golimumab in participants with active RA despite concurrent MTX therapy. Approximately 564 participants will be randomly allocated to 1 of 2 treatment groups in a 2:1 ratio ie, Group 1(approximately 376 participants will receive golimumab + MTX) and Group 2 (approximately 188 participants will receive MTX + placebo). Total duration of study for each participant is 112 weeks. Safety will be evaluated by assessment of adverse events, tuberculosis testing and blood testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis (RA) for at least 3 months prior to screening
* Have been treated with and tolerated methotrexate (MTX) at a dose of at least 15 mg/week for at least 3 months prior to screening, and have been on a stable MTX dose of 15 mg/week to 25 mg/week for at least 4 weeks prior to screening
* Have an active RA, as defined by disease activity with at least 6 swollen and 6 tender joints, at the time of screening and at baseline
* C-Reactive Protein greater than or equal to 1.0 mg/dL at screening
* No history of latent or active tuberculosis prior to screening

Exclusion Criteria:

* Other inflammatory diseases, including but not limited to psoriatic arthritis, ankylosing spondylitis, systemic lupus erythematosus, or lyme disease
* Treated with disease modifying agents (other than methotrexate)/systemic immunosuppressives (eg, D-penicillamine, hydroxychloroquine, chloroquine, oral or parenteral gold, sulfasalazine, leflunomide, azathioprine, cyclosporine, mycophenolate mofetil) during the 4 weeks prior to first administration of study agent
* Received intra-articular (in the joint), intramuscular (in the muscle), or intravenous corticosteroids, including adrenocorticotropic hormone, during the 4 weeks prior to first administration of study agent
* Known allergy to human immunoglobulin proteins or other components of golimumab
* Received any commercial or investigational anti-tumor necrosis factor alpha therapy such as but not exclusively infliximab, golimumab, adalimumab or etanercept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (88):
- United States (9):
  - Daytona Beach, Florida
  - Miami, Florida
  - Palm Harbor, Florida
  - Moline, Illinois
  - Wheaton, Maryland
  - Worcester, Massachusetts
  - Lincoln, Nebraska
  - Cincinnati, Ohio
  - Lubbock, Texas
- Argentina (6):
  - Buenos Aires
  - Córdoba
  - Rosario
  - San Juan
  - San Miguel de Tucumán
  - Santa Fe
- Australia (5):
  - Cairns
  - Maroochydore
  - Melbourne
  - Woodville
  - Woolloongabba
- Colombia (5):
  - Antioquia
  - Barranquilla
  - Bogotá
  - Cali Valley Del Cauca
  - Medellín
- Hungary (7):
  - Budapest
  - Debrecen
  - Eger
  - Győr
  - Gyula
  - Szombathely
  - Veszprém
- Lithuania (5):
  - Alytus
  - Kaunas
  - Klaipėda
  - Šiauliai
  - Vilnius
- Malaysia (9):
  - George Town
  - Ipoh
  - Johor Bahru
  - Kota Kinabalu
  - Kuantan
  - Kuching
  - Precinct 7
  - Selangor Darul Ehasan
  - Seremban
- Mexico (5):
  - Guadalajara
  - León
  - Mexico City
  - México
  - Monterrey
- New Zealand (3):
  - Auckland
  - Takapuna Auckland
  - Timaru
- Poland (12):
  - Bialystok
  - Bydgoszcz
  - Działdowo
  - Elblag
  - Katowice
  - Lublin
  - Poznan
  - Sopot
  - Szczecin
  - Warsaw
  - Wroclaw
  - Włoszczowa
- Russia (7):
  - Chelyabinsk
  - Krasnoyarsk
  - Moscow
  - Petrozavodsk
  - Saint Petersburg
  - Saratov
  - Yekaterinburg
- South Korea (6):
  - Anyang
  - Daegu
  - Daejeon
  - Incheon
  - Pusan
  - Seoul
- Ukraine (9):
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
  - Odesa
  - Simferopol
  - Ternopil
  - Vinnitsa
  - Zaporizhzhya

REFERENCES:
- [Derived] Husni ME, Deodhar A, Schwartzman S, Chakravarty SD, Hsia EC, Leu JH, Zhou Y, Lo KH, Kavanaugh A. Pooled safety results across phase 3 randomized trials of intravenous golimumab in rheumatoid arthritis, psoriatic arthritis, and ankylosing spondylitis. Arthritis Res Ther. 2022 Mar 21;24(1):73. doi: 10.1186/s13075-022-02753-6. PMID 35313978
- [Derived] Lee JB, Broadwell A, Fan Y, Hu C, Adedokun OJ, Chakravarty SD, Zhou H, Xu Z, Leu JH. Population Pharmacokinetic and Exposure-Response Model Simulations: Predicted Exposure and Efficacy for Maintenance Doses of Intravenous Golimumab Every 6 or 8 Weeks in Patients With Moderately to Severely Active Rheumatoid Arthritis. Clin Ther. 2022 Mar;44(3):457-464.e2. doi: 10.1016/j.clinthera.2022.01.015. Epub 2022 Feb 17. PMID 35183373
- [Derived] Tesser J, Kafka S, DeHoratius RJ, Xu S, Hsia EC, Turkiewicz A. Efficacy and safety of intravenous golimumab plus methotrexate in patients with rheumatoid arthritis aged < 65 years and those >/= 65 years of age. Arthritis Res Ther. 2019 Aug 20;21(1):190. doi: 10.1186/s13075-019-1968-x. PMID 31429794
- [Derived] Standish KA, Huang CC, Curran ME, Schork NJ. Comprehensive analysis of treatment response phenotypes in rheumatoid arthritis for pharmacogenetic studies. Arthritis Res Ther. 2017 May 12;19(1):90. doi: 10.1186/s13075-017-1299-8. PMID 28494788
- [Derived] Bingham CO 3rd, Mendelsohn AM, Kim L, Xu Z, Leu J, Han C, Lo KH, Westhovens R, Weinblatt ME; GO-FURTHER Investigators. Maintenance of Clinical and Radiographic Benefit With Intravenous Golimumab Therapy in Patients With Active Rheumatoid Arthritis Despite Methotrexate Therapy: Week-112 Efficacy and Safety Results of the Open-Label Long-Term Extension of a Phase III, Double-Blind, Randomized, Placebo-Controlled Trial. Arthritis Care Res (Hoboken). 2015 Dec;67(12):1627-36. doi: 10.1002/acr.22556. PMID 25623393
- [Derived] Bingham CO 3rd, Weinblatt M, Han C, Gathany TA, Kim L, Lo KH, Baker D, Mendelsohn A, Westhovens R. The effect of intravenous golimumab on health-related quality of life in rheumatoid arthritis: 24-week results of the phase III GO-FURTHER trial. J Rheumatol. 2014 Jun;41(6):1067-76. doi: 10.3899/jrheum.130864. Epub 2014 May 1. PMID 24786931
- [Derived] Weinblatt ME, Westhovens R, Mendelsohn AM, Kim L, Lo KH, Sheng S, Noonan L, Lu J, Xu Z, Leu J, Baker D, Bingham CO; GO-FURTHER investigators. Radiographic benefit and maintenance of clinical benefit with intravenous golimumab therapy in patients with active rheumatoid arthritis despite methotrexate therapy: results up to 1 year of the phase 3, randomised, multicentre, double blind, placebo controlled GO-FURTHER trial. Ann Rheum Dis. 2014 Dec;73(12):2152-9. doi: 10.1136/annrheumdis-2013-203742. Epub 2013 Sep 3. PMID 24001888

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of intravenous administration of Golimumab 2mg/kg + methotrexate (MTX) in patients with Active Rheumatoid Arthritis despite treatment with MTX therapy. It was conducted between 14 September 2009 and 08 February 2013 and recruited participants at 92 sites in 13 countries worldwide.
Pre-assignment Details: 592 participants were randomly allocated to 2 treatment arms. At Week 16 some participants in Placebo arm switched to Golimumab earlier than the rest at Week 24. Thus, the Adverse Events are presented based upon the time when participants began to receive Golimumab in the following manner: Golimumab from Day 0, from Week 16 and from Week 24.
Groups:
- Group I: Placebo + Methotrexate (MTX): Participants randomized to receive their stable dose of commercial MTX (between 15-25 mg/week) and placebo IV infusions at Weeks 0, 4, 12, 16, and 20. Participants will be crossed over to Golimumab 2 mg/kg at Week 24, and receive administrations at Weeks 24, 28 and q8 weeks thereafter up to Week 100. Subjects randomized to Group I (Placebo + MTX) will have the opportunity to enter early escape at Week 16 and initiate Golimumab 2 mg/kg infusions (Weeks 16, 20, and q8 weeks up to Week 100) if they demonstrate a < 10% improvement in both tender and swollen joint count.
- Group II: Golimumab 2 mg/kg + Methotrexate (MTX): Participants randomized to receive 2 mg/kg of Golimumab intravenously at Weeks 0, 4, and q8 weeks up to Week 100. Participants will be maintained on their stable dose of commercial MTX (between 15 and 25 mg/week) throughout the study. Participants will receive a placebo infusion at Week 16 and Week 24 to maintain the blind.
Period: Overall Study
Arm/Group | Group I: Placebo + Methotrexate (MTX) | Group II: Golimumab 2 mg/kg + Methotrexate (MTX)
Started | 197 | 395
Completed | 160 | 326
Not Completed | 37 | 69
Not completed — Lost to Follow-up | 0 | 3
Not completed — Death | 2 | 2
Not completed — Withdrawal by Subject | 15 | 16
Not completed — Lack of Efficacy | 5 | 7
Not completed — Adverse Event | 12 | 32
Not completed — Protocol Violation | 2 | 2
Not completed — Other | 1 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I: Placebo + Methotrexate (MTX) | Group II: Golimumab 2 mg/kg + Methotrexate (MTX) | Total
Number analyzed (Participants) | 197 | 395 | 592
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (11.26) | 51.9 (12.55) | 51.8 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 326 | 483
  Male | 40 | 69 | 109
Region of Enrollment [Number; unit: participants]
  Argentina | 28 | 54 | 82
  Australia | 3 | 6 | 9
  Columbia | 12 | 25 | 37
  Hungary | 10 | 21 | 31
  Korea, Republic of | 4 | 12 | 16
  Lithuania | 20 | 44 | 64
  Malaysia | 8 | 18 | 26
  Mexico | 13 | 25 | 38
  New Zealand | 2 | 4 | 6
  Poland | 36 | 65 | 101
  Russian Federation | 23 | 46 | 69
  Ukraine | 32 | 58 | 90
  United States | 6 | 17 | 23

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With an American College of Rheumatology (ACR) 20 Response at Week 14
Description: An ACR 20 response is defined as a greater than or equal to 20 percent improvement from baseline in: 1. Swollen (66 joints) and tender (68 joints) joint counts; 2. greater than or equal to 20 percentage improvement in at least 3 of the following 5 assessments: a. Participant's assessment of pain by Visual Analog Scale (VAS), (0 [no pain] to 10 [worst pain]) b. Participant's global assessment of disease activity by VAS c. Physician's global assessment of disease activity by VAS d. Participant's assessment of physical function as measured by the Health Assessment Questionnaire (HAQ) e. C-reactive protein.
Time Frame: Week 14
Population: Intent-to-treat: all patients analyzed according to the treatment for which they were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group I: Placebo + Methotrexate (MTX) | Group II: Golimumab 2 mg/kg + Methotrexate (MTX)
Number analyzed (Participants) | 197 | 395
Percentage of Participants | 24.9 | 58.5
Statistical Analysis 1: Comparison: Group I: Placebo + Methotrexate (MTX) vs Group II: Golimumab 2 mg/kg + Methotrexate (MTX); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Proportion of Participants With Moderate or Good Response in Disease Activity Index Score 28 (DAS28) Using C-reactive Protein (CRP) at Week 14
Description: DAS28 using CRP is an index to measure the disease activity in participants with rheumatoid arthritis combining tender joints (28 joints), swollen joints (28 joints), CRP, and participant's global assessment of disease activity. The DAS28 score ranges from 0 (best) to 10 (worst). DAS28 score above 5.1 means high disease activity whereas a DAS28 below 3.2 indicates low disease activity. Higher scores indicate worsening. A decrease in DAS28 score >1.2 is being referred to as a "good response" and a decrease of 0.6-1.2 as a "moderate response".
Time Frame: Week 14
Population: Intent-to-treat: all patients analyzed according to the treatment for which they were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group I: Placebo + Methotrexate (MTX) | Group II: Golimumab 2 mg/kg + Methotrexate (MTX)
Number analyzed (Participants) | 197 | 395
Percentage of Participants | 40.1 | 81.3
Statistical Analysis 1: Comparison: Group I: Placebo + Methotrexate (MTX) vs Group II: Golimumab 2 mg/kg + Methotrexate (MTX); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Score at Week 14
Description: The HAQ is 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0 (no difficulty), to 3 (inability to perform a task in that area). HAQscore on a scale ranges from 0 (no disability) to 3 (completely disabled). Higher scores indicate worsening.
Time Frame: Week 14
Population: Intent-to-treat: all patients analyzed according to the treatment for which they were randomized.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Group I: Placebo + Methotrexate (MTX) | Group II: Golimumab 2 mg/kg + Methotrexate (MTX)
Number analyzed (Participants) | 197 | 395
Scores on a scale | 0.1250 (0.55770) | 0.5000 (0.57706)
Statistical Analysis 1: Comparison: Group I: Placebo + Methotrexate (MTX) vs Group II: Golimumab 2 mg/kg + Methotrexate (MTX); Test type: Superiority or Other; p < 0.001, ANOVA of van der Waerden scores

4. Secondary Outcome: Proportion of Participants Who Achieved American College of Rheumatology (ACR) 50 Response at Week 24
Description: An ACR 50 response is defined as a greater than or equal to 50 percent improvement from baseline in: 1. Swollen (66 joints) and tender (68 joints) joint counts; 2. greater than or equal to 50 percentage improvement in 3 of the following 5 assessments: a. Participant's assessment of pain by Visual Analog Scale (VAS) (0-10 cm) b. Participant's global assessment of disease activity by VAS (0-10 cm) c. Physician's global assessment of disease activity by VAS (0-10 cm) d. Participant's assessment of physical function as measured by the Health Assessment Questionnaire (HAQ) e. C reactive protein.
Time Frame: Week 24
Population: Intent-to-treat: all patients analyzed according to the treatment for which they were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group I: Placebo + Methotrexate (MTX) | Group II: Golimumab 2 mg/kg + Methotrexate (MTX)
Number analyzed (Participants) | 197 | 395
Percentage of Participants | 13.2 | 34.9
Statistical Analysis 1: Comparison: Group I: Placebo + Methotrexate (MTX) vs Group II: Golimumab 2 mg/kg + Methotrexate (MTX); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

5. Secondary Outcome: Change From Baseline in Total Van Der Heijde Modified Sharp (vdH-S) Score at Week 24.
Description: Total vdH-S score is sum of joint erosion score and joint-space narrowing (JSN) score. Joint erosion score summarizes erosion severity in 32 joints of hands and 12 joints of feet. Each joint scored from 0 (no erosion) to 5 (extensive loss of bone from more than one half of the articulating bone). Maximal erosion score is 280. JSN score summarizes severity of JSN in 30 joints of hands and 12 joints of feet. Assessment of JSN, including subluxation, is scored from 0 (normal) to 4 (bony ankylosis or complete luxation). Maximal JSN score is 168. Thus, the worst possible vdH-S score is 448.
Time Frame: Week 24
Population: Intent-to-treat: all patients analyzed according to the treatment for which they were randomized.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Group I: Placebo + Methotrexate (MTX) | Group II: Golimumab 2 mg/kg + Methotrexate (MTX)
Number analyzed (Participants) | 197 | 395
Scores on a scale | 1.09 (3.194) | 0.03 (1.899)
Statistical Analysis 1: Comparison: Group I: Placebo + Methotrexate (MTX) vs Group II: Golimumab 2 mg/kg + Methotrexate (MTX); Test type: Superiority or Other; p < 0.001, ANOVA of van der Waerden scores

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for the duration of study (100 weeks) and follow-up (12 weeks).
Description: The total number of adverse events listed in the "Other (non-Serious) Adverse Events" table is based upon a cut-off of greater than or equal to 5 percent of patients experiencing the adverse event in any treatment arm.
Groups:
- Placebo + MTX -> Golimumab 2 mg/kg + MTX at Week 16: Participants received placebo only through Week 16 and met early escape criteria or subjects who received first placebo and later inadvertently received Golimumab prior or at Week 16. The follow-up period for this treatment group begins once a participant switches to Golimumab 2 mg/kg. Participants may have missed one or more study agent doses.
- Placebo + MTX -> Golimumab 2 mg/kg + MTX at Week 24: Participants received placebo only through Week 24 or subjects who received first placebo and later inadvertently received Golimumab after Week 16 through Week 24. The follow-up period for this treatment group begins once a participants switches to Golimumab 2 mg/kg. Participants may have missed one or more study agent doses.
- Golimumab 2 mg/kg + MTX: Participants were assigned to Golimumab 2 mg/kg + MTX and received at least one 2 mg/kg Golimumab. The follow-up period for this treatment group begins with the first dose of Golimumab 2 mg/kg. Participants may have missed one or more Golimumab doses.
- Combined Golimumab: Participants in the reporting groups: Placebo + MTX -> Golimumab 2 mg/kg + MTX at Week 16, Placebo + MTX -> Golimumab 2 mg/kg + MTX at Week 24, and Golimumab 2 mg/kg + MTX.
Arm/Group | Placebo + MTX -> Golimumab 2 mg/kg + MTX at Week 16 | Placebo + MTX -> Golimumab 2 mg/kg + MTX at Week 24 | Golimumab 2 mg/kg + MTX | Combined Golimumab
Serious Adverse Events (participants affected / at risk) | 11/68 | 17/121 | 78/395 | 106/584
Other Adverse Events (participants affected / at risk) | 34/68 | 38/121 | 199/395 | 271/584
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + MTX -> Golimumab 2 mg/kg + MTX at Week 16 (N=68) | Placebo + MTX -> Golimumab 2 mg/kg + MTX at Week 24 (N=121) | Golimumab 2 mg/kg + MTX (N=395) | Combined Golimumab (N=584)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 1 | 2
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 2
Cor pulmonale chronic (Cardiac disorders) | 0 | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 2 | 3
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Cyst (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Sudden death (General disorders) | 0 | 1 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 0 | 1 | 1
Endophthalmitis (Infections and infestations) | 1 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 2 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1
Infective spondylitis (Infections and infestations) | 0 | 0 | 1 | 1
Intervertebral discitis (Infections and infestations) | 0 | 0 | 1 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Lung abscess (Infections and infestations) | 0 | 0 | 1 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 4 | 5
Pneumonia cryptococcal (Infections and infestations) | 0 | 1 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Sepsis syndrome (Infections and infestations) | 0 | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 1
Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 1
Tuberculous pleurisy (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 3 | 4
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 10 | 12
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 1 | 2
Iiird nerve paresis (Nervous system disorders) | 0 | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 2 | 2
Lacunar infarction (Nervous system disorders) | 0 | 0 | 1 | 1
Radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 1
Nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 1
Bartholinitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Breast disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Arterial rupture (Vascular disorders) | 0 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + MTX -> Golimumab 2 mg/kg + MTX at Week 16 (N=68) | Placebo + MTX -> Golimumab 2 mg/kg + MTX at Week 24 (N=121) | Golimumab 2 mg/kg + MTX (N=395) | Combined Golimumab (N=584)
Bronchitis (Infections and infestations) | 6 | 9 | 37 | 52
Nasopharyngitis (Infections and infestations) | 3 | 8 | 28 | 39
Pharyngitis (Infections and infestations) | 0 | 7 | 26 | 33
Upper respiratory tract infection (Infections and infestations) | 5 | 8 | 54 | 67
Urinary tract infection (Infections and infestations) | 3 | 7 | 26 | 36
Alanine aminotransferase increased (Investigations) | 8 | 3 | 27 | 38
Aspartate aminotransferase increased (Investigations) | 5 | 2 | 18 | 25
Hepatic enzyme increased (Investigations) | 4 | 0 | 6 | 10
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 9 | 3 | 33 | 45
Headache (Nervous system disorders) | 5 | 2 | 27 | 34
Hypertension (Vascular disorders) | 8 | 4 | 27 | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less